CLINICAL TRIAL: NCT05817851
Title: Efficacy of Early Intravenous High-dose Vitamin C in Post-cardiac Arrest Shock: a Multicenter, Randomized Controled Trial.
Brief Title: Efficacy of Early Intravenous High-dose Vitamin C in Post-cardiac Arrest Shock.
Acronym: VICEPAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier de Bethune (Network)
Collaborators: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other); University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Ascorbic Acid; Thiamine

STUDY DESIGN:
Intervention Model Description: The study is a phase II multicenter prospective controlled open-label trial randomized in two parallel groups :
  * Expérimental group
  * Control group
  Patient number to be enrolled : 234, Study duration :24 months and 28 days, Inclusion duration : 24 months, Patient participation : duration : 28 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): - Control group (standard treatment): post-cardiac arrest care will be provided, including temperature control, according to current international guidelines and local procedures. Standard IV vit-C supplementation will be allowed for dosages up to 1000 mg a day from day 4 after randomization, as well as thiamin supplementation.
  Interventions: Drug: standard treatment
- Experimental group (Experimental): - Experimental group (IV high-dose vit-C): in addition of standard post-CA as the control group, patients will receive an IV high-dose vit-C 50mg/kg infusion every 6 hours, started within the hour after randomization, for 3 days. In addition, all patients will receive intravenous thiamine 200 mg twice a day for 3 days to limit the oxalate production.
  Interventions: Drug: Vitamin C (Laroscorbine) + Vitamin B1 (Bevitine)

INTERVENTIONS:
Drug: Vitamin C (Laroscorbine) + Vitamin B1 (Bevitine) — in addition of standard post-CA as the control group, patients will receive an IV high-dose vit-C 50mg/kg infusion every 6 hours, started within the hour after randomization, for 3 days. In addition, all patients will receive intravenous thiamine 200 mg twice a day for 3 days to limit the oxalate production.
  Other Names: Laroscorbine + Bevitine
  Arms: Experimental group
Drug: standard treatment — no intervention Standard IV vit-C supplementation will be allowed for dosages up to 1000 mg a day from day 4 after randomization, as well as thiamin supplementation.
  Arms: Control group

SUMMARY:
Among patients admitted after an out-of-hospital cardiac arrest (OHCA) in intensive care unit (ICU), almost two thirds of patients will develop in the first hours a post-cardiac arrest (CA) shock. This post-CA shock, combines cardiac and hemodynamic failure, generally resulting in multi-organ failure and early death in up to 35% of patients. Experimental data suggest that intravenous ascorbic acid (vitamin C) may attenuate inflammation and vascular injury related to sepsis or surgery. Preclinical and clinical studies also provide safety data of high dose intravenous vitamin C (> 200mg/kg/day) with no significant adverse event reported and favorable impact on outcome. Experimental data also suggest beneficial effect of vitamin C in post-CA management with improvement of shock and multi-organ failure with potential benefit on neuroprotection and outcome.

The study is a phase II multicenter prospective controlled open-label trial randomized in two parallel groups :

* Expérimental group: Standard of care care for post-CA shock + Vitamin C (Vit-C) 200mg/kg/d IV (started as early as possible, no later than 1 h after randomization + thiamin (Vit B1) 200mg every 12 h during 3 days.
* Control group: Standard of care care for post CA shock according international guidelines.

Patient number to be enrolled : 234, Study duration :24 months and 28 days, Inclusion duration : 24 months, Patient participation : duration : 28 days

ELIGIBILITY:
Inclusion Criteria:

* patients still comatose (Glasgow coma scale < 8) after an OHCA of presumed cardiac origin with ROSC < 60 min;
* and treated with a norepinephrin or an epinephrin continuous infusion during at least 30 min before randomization to maintain mean arterial pressure (MAP) ≥ 65 mmHg.

Exclusion Criteria:

* patients still comatose (Glasgow coma scale < 8) after an OHCA of presumed cardiac origin with ROSC < 60 min;
* and treated with a norepinephrin or an epinephrin continuous infusion ≥ 0.2µg/kg/h, within 4 hours after OHCA, during at least 30 min/h to maintain mean arterial pressure (MAP) ≥ 65 mmHg.

Exclusion criteria:

* minor or pregnant women;
* OHCA from evident extracardiac cause (trauma, bleeding, poisoning, etc.);
* interval between RACS and randomization > 6 hours;
* extracorporeal circulatory assistance requirement in the first 4 hours after OHCA;
* history of urolithiasis, oxalate nephropathy or hemochromatosis;
* glucose-6-phosphate deshydrogenase deficiency; nephrolithiasis, hyperoxalyurie
* patients already treated with vit-C; known vit-C deficit;
* inclusion in another study;
* pre-existent severe chronic kidney disease (glomerular filtration rate < 30ml/min);
* treatment limitationsor moribound
* Patient with derpived freedom or with legal protective measures.
* Patient not covered by French national health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01-24 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of weaning from vasopressors at day 3 after OHCA. | day 3
  Cumulative incidence of weaning from vasopressors at day 3 after OHCA.

SECONDARY OUTCOMES:
Cumulative incidence of death by refractory shock within 7 days after OHCA. | day 7 after OHCA
  Cumulative incidence of death by refractory shock within 7 days after OHCA.
the neurological outcome at day 28 after OHCA, with mRS range from 0 to 3. | day 28 after OHCA
  Assessed using the mRS (favorable neurological outcome will be considered if mRS range from 0 to 3; Unfavorable neurological outcome will be considered if mRS range from 4 to 6).
The maximal vasopressors infusion dose within 3 days after OHCA. | 72 hours after OHCA
  The maximal vasopressors infusion dose within 3 days after OHCA.
The delta SOFA (sepsis-related organ failure assessment score) is defined as the difference between SOFA admission and SOFA at 72 hours after OHCA. | 72 hours after OHCA
  Death within 72 hours will be counted as the maximum SOFA score (i.e. 24 points).
The lower arterial lactate level at day 3 after OHCA. | 72 hours after OHCA
  The lower arterial lactate level at day 3 after OHCA.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - CH d'Arras, Arras
  - Centre Hospitalier Béthune, Béthune
  - CHI Nord-Ardennes, Charleville-Mézières
  - Centre Hospitalier de Dieppe, Dieppe
  - GHEF Site Marne La Vallée, Jossigny
  - Centre Hospitalier de LENS, Lens
  - Centre Hospitalier Universitaire de LILLE, Lille
  - CH de Melun (GHSIF), Melun
  - Hôpital Lariboisière, Paris
  - Centre Hospitalier de Rouen, Rouen
  - Centre Hospitalier Toulon La Seyne sur Mer, Toulon
  - Centre Hospitalier de Valenciennes, Valenciennes
  - CH de Versailles, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chelly J, Peres N, Sboui G, Maizel J, Beuzelin M, Nigeon O, Preau S, Vong LVP, Tamion F, Lambiotte F, Deye N, Bertrand T, Behal H, Ducros L, Vinsonneau C. Early intravenous high-dose vitamin C in postcardiac arrest shock (VICEPAC): study protocol for a randomised, single-blind, open-label, multicentre, controlled trial. BMJ Open. 2024 Sep 24;14(9):e087303. doi: 10.1136/bmjopen-2024-087303. PMID 39317492